CLINICAL TRIAL: NCT04349280
Title: A Phase Ib Trial to Evaluate the Efficacy and Safety of Bintrafusp Alfa Monotherapy in Metastatic or Locally Advanced/Unresectable Urothelial Cancer With Disease Progression or Recurrence Following Treatment With a Platinum Agent
Brief Title: A Study to Evaluate the Efficacy and Safety of Bintrafusp Alfa (M7824) Monotherapy in Metastatic or Locally Advanced Urothelial Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Primary investigator withdrew the participant due to an SAE
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 213152
Record Dates: First submitted 2020-04-15; First posted 2020-04-16 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Neoplasms
Keywords: Bintrafusp Alfa; Platinum Agent; Response Evaluation Criteria in Solid Tumors; Urothelial Cancer; M7824
MeSH Terms: conditions — Neoplasms | interventions — bintrafusp alfa protein, human

STUDY DESIGN:
Intervention Model Description: This is a single arm study.
Masking Description: This is an open label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants receiving bintrafusp alfa (Experimental): Participants will receive bintrafusp alfa.
  Interventions: Drug: Bintrafusp alfa

INTERVENTIONS:
Drug: Bintrafusp alfa — Participants will receive bintrafusp alfa.

SUMMARY:
The purpose of this study is to evaluate bintrafusp alfa in participants with metastatic or locally advanced urothelial cancer. This trial provides the first evaluation of bintrafusp alfa in participants with urothelial cancer that has progressed following platinum therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants can give signed informed consent/assent.
* Participants with histologically confirmed locally advanced or metastatic or locally advanced/unresectable urothelial carcinoma (including renal, pelvis, ureter, urinary bladder, urethra).
* Able to provide, a tumor tissue sample collected during screening and prior to administration of bintrafusp alfa.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
* Participants with adequate organ system functions.
* Life expectancy of at least 12 weeks.
* A female is eligible if she is not pregnant or breastfeeding.

Exclusion Criteria:

* Active brain and/or leptomeningeal disease that is symptomatic or requires therapeutic intervention. Participants with asymptomatic central nervous system (CNS) metastases who are clinically stable as demonstrated by serial brain images and have no requirement for corticosteroids for at least 14 days prior to enrollment are eligible.
* History of malignancy other than urothelial cancer within the last 3 years except for localized tumors that have been treated with curative intent or have not required therapy in the past 2 years. (e.g., resected non-melanoma skin cancer).
* No more than 2 lines of systemic therapy for the treatment of metastastic disease. If the most recent therapy was not a platinum-based regimen, the participant must have progressed on or after that therapy.
* Cirrhosis or current unstable liver or biliary disease per investigator assessment.
* Current pneumonitis or history of non-infectious pneumonitis that required systemic immunosuppressive treatment.
* Active autoimmune disease that required systemic immunosuppressive treatment within the past 2 years.
* Received prior allogeneic/autologous bone marrow or solid organ transplant.
* Receiving systemic corticosteroids (>10 milligrams [mg] daily oral prednisone or equivalent) or other immunosuppressive agent within 7 days prior to study treatment. Inhaled or topical steroids are permitted.
* Known severe hypersensitivity reactions to monoclonal antibodies or any ingredient used in the study treatment formulation (Grade >=3 National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE] version 5.0).
* Active infection requiring systemic therapy.
* Received any live vaccine within 30 days prior first dose of intervention.
* Known history of positive test for human immunodeficiency virus (HIV) with the exception of participants with cluster of differentiation 4 (CD4) + T-cell (CD4+) counts >=350 cells per microliter (cells /uL) and no history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections.
* Active hepatitis B virus (HBV) (HBV surface antigen-positive).
* Active hepatitis C virus (HCV) infection, or positive HCV antibody, with the exception of participants that 1. Have HCV viral load below the limits of quantitation and 2. Completed curative antiviral therapy or are receiving and compliant with antiviral therapy.
* History or evidence of cardiac abnormalities within the 6 months prior to first dose of intervention.
* Participants with history of bleeding diathesis or recent major bleeding events considered by the Investigator as high risk for investigational drug treatment are also excluded.
* Any other serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the participant to receive protocol therapy, or interfere with the interpretation of study results.
* Received prior systemic anti-cancer therapy within 2 weeks prior to study treatment.
* Received prior therapy with an anti-programmed death 1 (PD-1), anti-programmed death Ligand 1 (anti-PD-L1), anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Received prior therapy targeting transforming growth factor (TGF) beta - (e.g., Galunistertib).
* Received radiation therapy (or other non-systemic disease therapy) within 2 weeks prior to study treatment.
* Undergone major surgery within 4 weeks prior to administration of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (2):
  - GSK Investigational Site, Lake Success, New York
  - GSK Investigational Site, Cincinnati, Ohio
- GSK Investigational Site, Toronto, Ontario, Canada
- France (4):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Villejuif
- GSK Investigational Site, Amsterdam, Netherlands
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Main Study - Bintrafusp Alfa: Participants with metastatic or locally advanced/unresectable urothelial cancer with disease progression or recurrence received intravenous (IV) infusion of 1200 milligram (mg) of bintrafusp alfa over 1 hour once every 2 weeks up to 79 weeks
- PACT Phase - Bintrafusp Alfa: Participants with metastatic or locally advanced/unresectable urothelial cancer with disease progression or recurrence received intravenous (IV) infusion of 1200 milligram (mg) of bintrafusp alfa over 1 hour once every 2 weeks up to approximately 56 weeks.
Period: Main Study (Up to Approx. 95 Weeks)
Arm/Group | Main Study - Bintrafusp Alfa | PACT Phase - Bintrafusp Alfa
Started | 25 | 0
Completed | 12 | 0
Not Completed | 13 | 0
Not completed — Ongoing | 1 | 0
Not completed — Death | 12 | 0
Period: PACT Phase (Up to Approx. 56 Weeks)
Arm/Group | Main Study - Bintrafusp Alfa | PACT Phase - Bintrafusp Alfa
Started | 0 | 1 (Participants who were ongoing in the main study entered PACT Phase.)
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Main Study - Bintrafusp Alfa
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.3 (7.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Overall Response Rate (ORR) Assessed by Investigator Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Confirmed overall response rate (ORR) defined as the percentage of participants with a confirmed complete response (CR) or confirmed partial response (PR) via investigator assessment per RECIST (Response Evaluation Criteria In Solid Tumors Criteria) v1.1 relative to the total number of participants in the analysis population. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm).
Time Frame: Up to approximately 22 months
Population: Safety population included all participants who were administered at least 1 infusion of bintrafusp alfa.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Main Study - Bintrafusp Alfa
Number analyzed (Participants) | 25
Percentage of Participants | 20.0 [6.83 to 40.70]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Treatment Emergent Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether considered related to the study intervention. A SAE is defined as any untoward medical occurrence that, at any dose is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity and is a congenital anomaly/birth defect. AEs which start or worsen on or after Bintrafusp alfa infusion are defined as treatment-emergent.
Time Frame: Up to approximately 22 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Bintrafusp Alfa
Number analyzed (Participants) | 25
Participants
  Treatment Emergent AEs | 25
  Treatment Emergent SAEs | 17

3. Secondary Outcome: Number of Participants With Worst Grade Treatment Emergent AEs
Description: Treatment emergent adverse events were analyzed using National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0. Graded from Grade 1: mild asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated, Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL), Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL, Grade 4: Life-threatening consequences; urgent intervention indicated, Grade 5: death related AE. Higher grade indicates more severe condition. AEs which start or worsen on or after Bintrafusp alfa infusion are defined as treatment-emergent.
Time Frame: Up to approximately 22 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study - Bintrafusp Alfa
Number analyzed (Participants) | 25
Participants
  Grade 1 | 1
  Grade 2 | 6
  Grade 3 | 15
  Grade 4 | 1
  Grade 5 | 2

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to approximately 95 weeks for main study and up to approximately 56 weeks for PACT phase.
Description: Safety population included all participants who were administered at least 1 infusion of bintrafusp alfa.
Arm/Group | Main Study - Bintrafusp Alfa | PACT Phase - Bintrafusp Alfa
All-Cause Mortality (participants affected / at risk) | 12/25 | 0/1
Serious Adverse Events (participants affected / at risk) | 17/25 | 1/1
Other Adverse Events (participants affected / at risk) | 21/25 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study - Bintrafusp Alfa (N=25) | PACT Phase - Bintrafusp Alfa (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study - Bintrafusp Alfa (N=25) | PACT Phase - Bintrafusp Alfa (N=1)
Anaemia (Blood and lymphatic system disorders) | 11 (28) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (8) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (11) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (5) | 0 (0)
Asthenia (General disorders) | 5 (8) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 6 (8) | 0 (0)
Mucosal inflammation (General disorders) | 4 (5) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (5) | 0 (0)
Blood creatinine increased (Investigations) | 3 (4) | 0 (0)
Cell death (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (6) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (4) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (17) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/80/NCT04349280/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT04349280/SAP_001.pdf